CLINICAL TRIAL: NCT02856425
Title: Phase Ib Trial Of Pembrolizumab And Nintedanib
Brief Title: Trial Of Pembrolizumab And Nintedanib
Acronym: PEMBIB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004511-21; 2015/2329 (Other: CSET Number)
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Patients With Any Advanced Solid Tumors
MeSH Terms: interventions — nintedanib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Colorectal adenocarcinoma (not mismatch repair deficient by either PCR and/or IHC) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Gastric or gastroesophageal adenocarcinoma (not mismatch repair deficient by either PCR and/or IHC (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Urothelial cancer (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Renal Cell cancer (RCC) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Mesothelioma (MPM) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Cervical Cancer (CC) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Hepatocellular (HCC) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Thymic Carcinoma (TC) (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab
- Patients with advanced cancers and high tumor mutational burden (TMB-High) (Experimental): High tumor mutational burden (TMB-High) on their circulating tumor DNA (ctDNA) as defined by more than twenty mutations per megabase (≥20Mut/Mb) on FoundationOne Liquid CDx assay
  Interventions: Drug: Nintedanib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nintedanib — Nintedanib oral tablets. An angiokinase inhibitor targeting VEGFR 1-3, FGFR 1-3, and PDGFR α/β as well as RET. Refer to current IB for product details
Drug: Pembrolizumab — Pembrolizumab, Intravenous. An IgG4 anti-PD-1 blocking monoclonal antibody. Refer to current IB for product details

SUMMARY:
Both anti-angiogenesis and anti PD1 immunotherapy have shown beneficial efficacy in solid tumors and in particular in NSCLC. Therefore it is of interest to investigate whether the combination of these two approaches is tolerable. Moreover, comprehensive pre-clinical and clinical rationale sustain the hypothesis that anti-VEGF could synergize with immunotherapy for the benefit of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patients with advanced/metastatic cancer who have progressed after at least one line of standard therapy or are intolerant to standard therapy. Patients must fit into one of the following groups:

   Colorectal adenocarcinoma (not mismatch repair deficient by either PCR and/or IHC) Gastric or gastroesophageal adenocarcinoma (not mismatch repair deficient by either PCR and/or IHC Patients with advanced or metastatic Urothelial cancer (UC) Patients with advanced Renal Cell cancer (RCC) Patients with advanced Mesothelioma (MPM) Patients with advanced squamous cell carcinoma in Cervical Cancer (CC) Patients with advanced Hepatocellular (HCC) Patients with advanced Thymic Carcinoma (TC) Patients with advanced cancers and high tumor mutational burden (TMB-High) on their circulating tumor DNA (ctDNA) as defined by more than twenty mutations per megabase (≥20Mut/Mb) on FoundationOne Liquid CDx assay. Patients should be without known therapeutic options to provide clinical benefit.
3. ECOG performance status of score 0 or 1
4. Adequate organ function as defined by the following criteria :

   * Proteinuria ≤ Grade 2 NCI CTCAE v4.03
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥ 40 mL/min
   * Total bilirubin within normal range (≤ 1.5 x ULN if HCC)
   * AST and ALT ≤ 1.5 x upper limit of normal (ULN); if liver metastases AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN if HCC)
   * Coagulation parameter : International normalized ratio (INR) < 2, prothrombin time (PT) and partial thromboplastin time (PTT) < 50% of deviation of ULN
   * Absolute Neutrophils count (ANC) ≥ 1000 cells/mm^3
   * Platelets ≥100 000 cells/mm^3
   * Hemoglobin ≥ 9.0 g/dL
5. At least one measurable lesion according to RECIST v1.1 (Appendix 4) criteria and modified RECIST for mesothelioma only (Appendix 6) or any other baseline prerequisite for the assessment of the principal judgment criteria.
6. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment. Both sexually active females and males (and their female partners) patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 4 months after last study drug administration.
7. Signed and dated written informed consent prior to admission to the study
8. Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

1. Prior treatment with nintedanib
2. Known hypersensitivity to trial drugs or their excipients, peanut or soya or to contrast media
3. Prior treatment with pembrolizumab or any other anti PD1 or anti-PDL1 agents
4. Concurrent steroid medication (except topical or aerosol steroids). Any steroid medication should have been stopped for more than 7 days prior beginning of therapy.
5. History of autoimmune/immune mediated inflammatory disease, including but not limited to colitis, pneumonitis, hepatitis, hypophysitis, nephritis, hyperthyroidism, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, vasculitis, or glomerulonephritis (see Appendix 3). Patients with a history of auto-immune endocrinopathy (hypo/hyper thyroiditis, type 1 diabetes mellitus, …) and who are stable on hormone replacement therapy are eligible for the study. Patients with a history of vitiligo, pelade, cutaneous psoriasis and grade 1-2 Sjogren syndrome are eligible.
6. Chemo-, hormono-, radio- (except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks or 5 half-life times (whatever the shortest) prior to treatment with the trial drugs.
7. Administration of a live, attenuated vaccine within 4 weeks before registration
8. Treatment with systemic immunosuppressive medications (including but not limited to steroids azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to registration
9. Radiotherapy to the target lesion (unless a progression after radiotherapy has been documented)
10. Persistence of clinically relevant treatment-related toxicity from previous chemotherapy, targeted therapy and/or radiotherapy
11. Active brain metastases or leptomeningeal disease. Clinically asymptomatic brain metastases and clinically asymptomatic leptomeningeal disease are allowed (treatment with steroids prior initiation of the trial is not allowed). Patients with Diffuse Intrinsic Pontine Gliomas, even asymptomatic, are not allowed.
12. Radiographic evidence of cavitary tumors with local invasion of major blood vessels and/or at risk for perforation
13. History of clinically significant hemoptysis within the past 3 months (more than one teaspoon of fresh blood per day)
14. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
15. Therapeutic anticoagulation with drugs requiring INR monitoring (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day)
16. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
17. History of clinically significant hemorrhagic or thromboembolic event in the past 6 months
18. Known inherited (genetic) predisposition to bleeding or thrombosis (such deficit in protein C/S) or acquired predisposition to thrombosis (such as anti-phospholipid syndromes)
19. History of significant cardiovascular diseases ( i.e. supraventricular tachycardia, uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
20. Ongoing uncontrolled auto-immune thyroiditis. Ancient thyroiditis currently stable with substitutive therapy should not be excluded from the trial.
21. Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix. A history of more than 3 years of local prostate cancer treated by surgery and without PSA elevation since surgery, or local breast carcinoma treated by surgery without relapse are eligible.
22. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
23. Known to be human immunodeficiency virus (HIV) positive;
24. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
25. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
26. Pregnancy or breast feeding,
27. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
28. Active alcohol or drug abuse
29. Intake of Ganoderma Lucidum mushroom and/or herbal remedies and/or traditional medicines within the past 4 weeks prior to start of study treatment or concomitantly with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
MTD of Nintedanib | Assessed within 24 months after study start
  The primary endpoint is to determine the MTD of nintedanib based on the assessment of DLT occurrence during treatment Course 1.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Marabelle, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (5):
- France (5):
  - Gustave Roussy, Villejuif, Val De Marne
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hôpital Bichat, Paris
  - IUCT--O, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baldini C, Danlos FX, Varga A, Texier M, Halse H, Mouraud S, Cassard L, Champiat S, Signolle N, Vuagnat P, Martin-Romano P, Michot JM, Bahleda R, Gazzah A, Boselli L, Bredel D, Grivel J, Mohamed-Djalim C, Escriou G, Grynszpan L, Bigorgne A, Rafie S, Abbassi A, Ribrag V, Postel-Vinay S, Hollebecque A, Susini S, Farhane S, Lacroix L, Parpaleix A, Laghouati S, Zitvogel L, Adam J, Chaput N, Soria JC, Massard C, Marabelle A. Safety, recommended dose, efficacy and immune correlates for nintedanib in combination with pembrolizumab in patients with advanced cancers. J Exp Clin Cancer Res. 2022 Jul 7;41(1):217. doi: 10.1186/s13046-022-02423-0. PMID 35794623